CLINICAL TRIAL: NCT04246957
Title: Quality of Life Comparison in Patients With Different Types of Alopecia
Acronym: RDACCQV
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2019_843_0001
Record Dates: First submitted 2020-01-21; First posted 2020-01-29 (Actual); Last update posted 2020-12-02 (Actual); Status verified 2020-12

CONDITIONS: Alopecia; Quality of Life
Keywords: alopecia; quality of life; partner
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: general quality of life questionary — Every patient will have to fill out a general quality of life questionary : DLQI (Dermatology Life Quality Index)
Behavioral: specific quality of life questionary — Every patient will have to fill out a specific quality of life questionary : Hair Specific Skindex 29.

SUMMARY:
Hair loss is a frequent cause of patient consultation in dermatology. It is known to have a strong impact on patients' quality of life for many reasons; such as esthetic aspect, financial implications, social consequences. Numerous studies have assessed the impact of some types of alopecia on patients' quality of life. One study compared the quality of life in patients with scarring alopecia with patients of non-scarring alopecia. No studies have compared quality of life between the different types of scarring alopecia nor different types of non-scarring alopecia. However, none have assessed the impact on the patient partner quality of life. In addition, few treatments for alopecia are covered by national health insurance in France. The main objective is to compare the impact on the quality of life in different types of alopecia. By using the average scores of the questionnaire Dermatology Life Quality Index (DLQI) for each type of alopecia.

ELIGIBILITY:
Inclusion Criteria:

* patients affiliated to social security
* patients able to understand and fill out a questionnaire
* patients over 18 years old
* patient consulting in the dermatology department of Amiens University Hospital for a primary alopecia

Exclusion Criteria:

* minors
* patients under guardianship, deprived of liberty
* scalp affections other than alopecia
* secondary alopecia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Every patient consulting in the dermatology department of Amiens' University Hospital for a primary alopecia will have to fill out 2 questionnaires of quality of life: one general (DLQI : Dermatology Life Quality Index) and one specific (Hair Specific Skindex 29). Every patient partner will have to complete one questionnaire of quality of life: FDLQI (Family DLQI).
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2019-03-04 (Actual); Primary Completion 2020-11-16 (Actual); Study Completion 2020-11-16 (Actual)

PRIMARY OUTCOMES:
Variation of score of questionnaire Dermatology Life Quality Index (DLQI) according alopecia type in patient life | at day 0
  The Dermatology life Quality Index (DLQI) is a ten-question questionnaire used to measure the impact of skin disease on the quality of life of an affected person. It is designed for people aged 16 years and above. There are 10 questions, covering the following topics: symptoms, embarrassment, shopping and home care, clothes, social and leisure, sport, work or study, close relationships, sex, treatment. Each question refers to the impact of the skin disease on the patient's life over the previous week. Each question is scored from 0 to 3, giving a possible score range form 0 (meaning no impact of skin disease on quality of life) to 30 (meaning maximum impact on quality of life).

SECONDARY OUTCOMES:
Variation of score of questionnaire Dermatology Life Quality Index (DLQI) according alopecia type in spouse life | at day 0
  The Dermatology life Quality Index (DLQI) is a ten-question questionnaire used to measure the impact of skin disease on the quality of life of an affected person. It is designed for people aged 16 years and above. There are 10 questions, covering the following topics: symptoms, embarrassment, shopping and home care, clothes, social and leisure, sport, work or study, close relationships, sex, treatment. Each question refers to the impact of the skin disease on the patient's life over the previous week. Each question is scored from 0 to 3, giving a possible score range form 0 (meaning no impact of skin disease on quality of life) to 30 (meaning maximum impact on quality of life).

CONTACTS AND LOCATIONS:
Overall Officials: Catherine LOK, Pr, Principal Investigator — CHU Amiens; Thomas Baltazard, MD, Principal Investigator — CHU Amiens; Nesrine Zitouni, MD, Principal Investigator — CHU Amiens; Fanny Dessirier, MD, Principal Investigator — CHU Amiens
Locations (1):
- CHU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No